CLINICAL TRIAL: NCT02106975
Title: Vitamin C Infusion for Treatment in Sepsis Induced Acute Lung Injury
Acronym: CITRIS-ALI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20000917; 1UM1HL116885-01 (NIH)
Record Dates: First submitted 2014-03-27; First posted 2014-04-08 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Acute Lung Injury; Sepsis
MeSH Terms: conditions — Acute Lung Injury; Sepsis | interventions — Ascorbic Acid; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ascorbic Acid (Active Comparator): 200mg/kg/day divided over 4 doses. Administered every 6 hours for 96 hours
  Interventions: Drug: Ascorbic Acid
- 5% Dextrose in Water (Placebo Comparator): 50ml every 6 hours for 96 hours
  Interventions: Drug: Placebo: 5% Dextrose in water

INTERVENTIONS:
Drug: Ascorbic Acid — Intervention
  Other Names: Vitamin C
  Arms: Ascorbic Acid
Drug: Placebo: 5% Dextrose in water — Placebo
  Arms: 5% Dextrose in Water

SUMMARY:
Hypothesis 1A: Vitamin C infusion will significantly attenuate sepsis-induced systemic organ failure as measured by Sequential Organ Failure Assessment (SOFA) score,

Hypothesis 1B: Vitamin C infusion will attenuate sepsis-induced lung injury as assessed by the oxygenation index and the VE40

Hypothesis 1C: Vitamin C infusion will attenuate biomarkers of inflammation (C-Reactive Protein, Procalcitonin), vascular injury (Thrombomodulin, Angiopoietin-2), alveolar epithelial injury (Receptor for Advanced Glycation Products), while inducing the onset of a fibrinolytic state (Tissue Factor Pathway Inhibitor).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have suspected or proven infection, and meet 2 out of 4 of the criteria for Systemic Inflammatory Response (SIRS) due to infection, and be accompanied by at least 1 criterion for sepsis-induced organ dysfunction, and meet all 5 criteria for Acute Respiratory Distress Syndrome (ARDS).
* Suspected or proven infection: (e.g., thorax, urinary tract, abdomen, skin, sinuses, central venous catheters, and central nervous system, see Appendix A).
* The presence of a systemic inflammatory response: Defined as: fever: >38ºC (any route) or hypothermia: <36ºC (core temp only), tachycardia: heart rate > 90 beats/min or receiving medications that slow heart rate or paced rhythm, leukocytosis: >12,000 WBC/µL or leukopenia: <4,000 WBC/µL or >10% band forms. Respiratory rate > 20 breaths per minute or PaCO2 < 32 or invasive mechanical ventilation.
* The presence of sepsis associated organ dysfunction: (any of the following thought to be due to infection)
* Sepsis associated hypotension (systolic blood pressure (SBP) < 90 mm Hg or an SBP decrease > 40 mm Hg unexplained by other causes or use of vasopressors for blood pressure support (epinephrine, norepinephrine, dopamine =/> 5mcg, phenylephrine, vasopressin)
* Arterial hypoxemia (PaO2/FiO2 < 300) or supplemental O2 > 6LPM.
* Lactate > upper limits of normal laboratory results
* Urine output < 0.5 ml/kg/hour for > two hours despite adequate fluid resuscitation
* Platelet count < 100,000 per mcL
* Coagulopathy (INR > 1.5)
* Bilirubin > 2 mg/dL
* Glasgow Coma Scale < 11 or a positive CAM ICU score
* ARDS characterized by all the following criteria
* Lung injury of acute onset, within 1 week of an apparent clinical insult and with progression of respiratory symptoms
* Bilateral opacities on chest imaging not explained by other pulmonary pathology (e.g. pleural effusions, lung collapse, or nodules)
* Respiratory failure not explained by heart failure or volume overload
* Decreased arterial PaO2/FiO2 ratio ≤ 300 mm Hg
* Minimum PEEP of 5 cmH2O (may be delivered noninvasively with CPAP to diagnose mild ARDS

Exclusion Criteria:

* Known allergy to Vitamin C
* inability to obtain consent;
* age < 18 years;
* No indwelling venous or arterial catheter in patients requiring insulin in a manner that requires glucose being checked more than twice daily (e.g. continuous infusion, sliding scale);
* presence of diabetic ketoacidosis;
* more than 48 hrs since meeting ARDS criteria;
* patient or surrogate or physician not committed to full support (not excluded if patient would receive all supportive care except for cardiac resuscitation);
* pregnancy or breast feeding,
* moribund patient not expected to survive 24 hours;
* home mechanical ventilation (via tracheotomy or noninvasive) except for CPAP/BIPAP used only for sleep-disordered breathing;
* home O2 > 2LPM, except for with CPAP/BIPAP
* diffuse alveolar hemorrhage (vasculitis);
* interstitial lung disease requiring continuous home oxygen therapy;
* Active kidney stone
* Non English speaking;
* Ward of the state (inmate, other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-04; Primary Completion 2017-11-16 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alpha B. Fowler, MD, Principal Investigator — Virginia Commonwealth University
Locations (5):
- United States (5):
  - Emory University and Grady Memorial Hospital, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - The Cleveland Clinic, Cleveland, Ohio
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fowler AA 3rd, Truwit JD, Hite RD, Morris PE, DeWilde C, Priday A, Fisher B, Thacker LR 2nd, Natarajan R, Brophy DF, Sculthorpe R, Nanchal R, Syed A, Sturgill J, Martin GS, Sevransky J, Kashiouris M, Hamman S, Egan KF, Hastings A, Spencer W, Tench S, Mehkri O, Bindas J, Duggal A, Graf J, Zellner S, Yanny L, McPolin C, Hollrith T, Kramer D, Ojielo C, Damm T, Cassity E, Wieliczko A, Halquist M. Effect of Vitamin C Infusion on Organ Failure and Biomarkers of Inflammation and Vascular Injury in Patients With Sepsis and Severe Acute Respiratory Failure: The CITRIS-ALI Randomized Clinical Trial. JAMA. 2019 Oct 1;322(13):1261-1270. doi: 10.1001/jama.2019.11825. PMID 31573637

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Started | 84 | 83
Completed | 59 | 44
Not Completed | 25 | 39
Not completed — Death | 25 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ascorbic Acid | 5% Dextrose in Water | Total
Number analyzed (Participants) | 84 | 83 | 167
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [39 to 67] | 57 [44 to 70] | 56 [41 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 45 | 45 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 82 | 81 | 163
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 13 | 19 | 32
  White | 68 | 60 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 84 | 83 | 167

OUTCOME MEASURES:

1. Primary Outcome: Modified Change in Sequential Organ Failure Assessment (mSOFA) Score
Description: mSOFA is a single score based on patient status of five different biological systems: respiratory, cardiovascular, coagulation, renal, and neurological. Scores range from 0 to 20 with higher scores indicated worse status.
Time Frame: 96 hours
Population: 3 participants were omitted from the analysis because the etiology of the patients SEPSIS was not representative of the typical SEPSIS patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
score on a scale | -2.96 (4.20) | -3.20 (3.30)

2. Primary Outcome: C-Reactive Protein at Study Hours 0, 48, 96, 168 When Compared to Placebo
Time Frame: up to 168 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
µg/ml
  0 hours | 109 (76) | 119 (67)
  48 hours | 80 (66) | 84 (52)
  96 hours | 56 (51) | 59 (52)
  168 hours | 54 (48) | 46 (33)

3. Primary Outcome: Thrombomodulin Protein at Study Hours 0, 48, 96, 168 When Compared to Placebo
Time Frame: Up to 168 hours
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
ng/ml
  0 hours | 14 (11) | 14 (8)
  48 hours | 15 (11) | 15 (10)
  96 hours | 15 (10) | 15 (10)
  168 hours | 14 (9) | 14 (9)

4. Secondary Outcome: Oxygenation Index (FiO2 x Mean Airway Pressure/PaO2) at Study Hour 0, 48, 96, 168 if Still Intubated in Ascorbate Infused Patient Compared to Placebo.
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
Index
  0 hour | 11 (10) | 10 (6)
  48 hours | 7 (5) | 7 (5)
  96 hours | 9 (6) | 7 (8)
  168 hours | 8 (8) | 8 (6)

5. Secondary Outcome: VE-40 (Vent RR x TV/Weight) x (PaCO2/40) at Study Hour 0, 48, 96, 168 if Still Intubated, in Ascorbate Infused Patient Compared to Placebo
Description: Estimate of Shunt
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmMercury
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
mmMercury
  0 hour | 127 (58) | 121 (60)
  48 hours | 127 (63) | 123 (51)
  96 hours | 127 (47) | 114 (46)
  168 hours | 115 (54) | 131 (77)

6. Secondary Outcome: mSOFA Scores at Hours 0, 48, 96
Description: as for outcome 1
Time Frame: Up to hour 96
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
units on a scale
  0 hours | 10 [7 to 12] | 10 [8 to 12]
  48 hours | 9 [5 to 12] | 8 [6 to 12]
  96 hours | 6 [4 to 10] | 6 [5 to 10]

7. Secondary Outcome: Ascorbate Level at Hour 0, 48, 96, 168
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
µM
  0 hour | 25 (18) | 26 (19)
  48 hours | 301 (355) | 24 (16)
  96 hours | 397 (580) | 26 (18)
  168 hours | 90 (145) | 28 (19)

8. Secondary Outcome: Ventilator Free Days to Day 28
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
days | 13 (11) | 11 (11)

9. Secondary Outcome: ICU-free Days at Day 28
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
days | 11 (10) | 8 (9)

10. Secondary Outcome: All Cause Mortality to Day 28
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
percentage of participants | 30 | 46

11. Secondary Outcome: Hospital-free Days at Day 60
Time Frame: Up to Day 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
days | 23 (22) | 15 (21)

12. Secondary Outcome: Procalcitonin at Study Hour 0, 48, 96, 168
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
ng/ml
  0 hour | 12 (23) | 27 (69)
  48 hours | 7 (18) | 9 (20)
  96 hours | 3 (6) | 4 (9)
  168 hours | 2 (3) | 3 (11)

13. Secondary Outcome: Receptor for Advanced Glycation Endpoints at Study Hour 0, 48, 96, 168
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
ng/ml
  0 hour | 6 (5) | 7 (5)
  48 hours | 4 (4) | 4 (3)
  96 hours | 4 (3) | 3 (2)
  168 hours | 3 (2) | 2 (2)

14. Secondary Outcome: Tissue Factor Pathway Inhibitor at Study Hour 0, 48, 96, 168
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
ng/ml
  0 hour | 46 (35) | 43 (28)
  48 hours | 42 (31) | 42 (33)
  96 hours | 42 (27) | 44 (28)
  168 hours | 44 (34) | 42 (31)

15. Secondary Outcome: Oxygenation Score: Pressure
Description: Oxygenation as measure by the ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2). Scores range from 100 to 300 with lower values indicating more worse outcomes
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Mercury
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
mm Mercury
  0 hour | 189 (96) | 214 (183)
  48 hours | 233 (115) | 246 (105)
  96 hours | 226 (109) | 244 (122)
  168 hours | 233 (134) | 254 (145)

16. Secondary Outcome: Oxygenation Score: Saturation
Description: Oxygenation as measure by the ratio of arterial oxygen saturation to fraction of inspired oxygen SpO2/FiO2
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
Ratio
  0 hour | 168 (51) | 177 (106)
  48 hours | 231 (81) | 220 (75)
  96 hours | 250 (101) | 244 (88)
  168 hours | 268 (107) | 299 (115)

17. Secondary Outcome: Coagulation
Description: Coagulation as measured by Platelets per unit of blood. Scores range from less than 20 to more than 150. Lower scores indicate worse outcomes
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Platelets/uL of Blood
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
Platelets/uL of Blood
  0 hour | 173 (123) | 175 (142)
  48 hours | 171 (133) | 147 (115)
  96 hours | 182 (141) | 165 (119)
  168 hours | 226 (180) | 228 (127)

18. Secondary Outcome: Liver Function
Description: Liver function as measured by Total Bilirubin. Normal levels range from 0.2 - 1.2. Levels greater than 1.2 indicate worse outcomes
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Median (Full Range); unit: Mg/dL
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
Mg/dL
  0 hour | 1 [0 to 22] | 1 [0 to 24]
  48 hours | 1 [0 to 23] | 1 [0 to 20]
  96 hours | 1 [0 to 22] | 1 [0 to 18]
  168 hours | 1 [0 to 28] | 1 [0 to 21]

19. Secondary Outcome: Cardiovascular Function
Description: Cardiovascular function as measured by Mean arterial pressure. Scores less than 70 mmHg indicate worse outcomes.
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
mmHg
  0 hour | 73 (13) | 73 (10)
  48 hours | 78 (15) | 79 (14)
  96 hours | 84 (16) | 84 (16)
  168 hours | 81 (14) | 83 (17)

20. Secondary Outcome: State of Consciousness
Description: State of consciousness as measure by Glasgow Coma Scale which gives a score based on eye, verbal, and motor responses. Scores range from 3 to 15 with lower scores indicating worse outcome
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
units on a scale
  0 hour | 8 [2 to 15] | 7 [3 to 15]
  48 hours | 9 [3 to 15] | 9 [3 to 15]
  96 hours | 10 [3 to 15] | 10 [3 to 15]
  168 hours | 10 [3 to 15] | 12 [3 to 15]

21. Secondary Outcome: Renal Function
Description: Renal function as measured by Creatinine. Scores range from less than 1.2 to greater than 5.0 with higher scores indicating worse outcomes
Time Frame: Up to hour 168
Population: as for outcome 1
Measure: Median (Full Range); unit: Mg/dL
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
Number analyzed (Participants) | 84 | 83
Mg/dL
  0 hour | 1 [0 to 6] | 2 [0 to 7]
  48 hours | 2 [0 to 8] | 1 [0 to 6]
  96 hours | 1 [0 to 7] | 1 [0 to 5]
  168 hours | 1 [0 to 7] | 1 [0 to 6]

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected for all days in the ICU, up to 4 days
Description: Due to the high level of adverse events normally associated with patients experiencing Sepsis Induced Acute Lung Injury, other than mortality, only drug related adverse events were tracked.
Arm/Group | Ascorbic Acid | 5% Dextrose in Water
All-Cause Mortality (participants affected / at risk) | 25/84 | 38/83
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/83
Other Adverse Events (participants affected / at risk) | 0/84 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT02106975/Prot_SAP_000.pdf